CLINICAL TRIAL: NCT00033072
Title: Assessment of Potential Interactions Between Intravenous Methamphetamine and Oral Selegiline
Brief Title: Assessment of Potential Interactions Between Methamphetamine and Selegiline - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: NIDA-CTO-0004-1; NCT00024882 (obsolete NCT alias)
Record Dates: First submitted 2002-04-05; First posted 2002-04-08 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2003-11

CONDITIONS: Amphetamine-Related Disorders
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — Selegiline

INTERVENTIONS:
Drug: Selegiline

SUMMARY:
The purpose of this study is to assess the potential interactions between intravenous methamphetamine and oral selegiline.

DETAILED DESCRIPTION:
To determine the safety of the selegiline concurrent with d-methamphetamine challenges of 15mg & 30mg i.v. with the focus being on cardiovascular responses (HR,BP) to the i.v. methamphetamine challenges. This is a randomized, single-blind, placebo-controlled, two-arm study design to evaluate the safety of selegiline treatment, compared to placebo treatment, concurrent with i.v. methamphetamine challenges.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers who meet DSM-4 criteria for methamphetamine abuse or dependence; non-treatment seeking individuals
* Be able to verbalize understanding of consent form; provide written informed consent

Exclusion Criteria:

* Please contact site for more information

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16
Dates: Start 2001-09; Study Completion 2002-10

PRIMARY OUTCOMES:
safety of selegiline
pharmacokinetic assessment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Newton, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Integrated Substance Abuse Program, Los Angeles, California, United States